CLINICAL TRIAL: NCT02664272
Title: Intraoperative Case Series Study: Trial Rasp Position Versus SL-PLUS™ MIA Ti/HA Femoral Hip Stem Position
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: SL MIA rasp 15-4567-03
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Total Hip Arthroplasty

SUMMARY:
A prospective, multicenter, observational study using the SL-PLUS™ MIA Ti/HA femoral hip stem with the appropriate set of instruments.

DETAILED DESCRIPTION:
The study objective was to evaluate if there was a difference between the femoral position of the last trial rasp and the final implant position of the SL-PLUS™ MIA Ti/HA femoral hip stem. The femoral position of rasp or stem was considered as the height of the implant / rasp in cranio-caudal direction.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* requires primary THA with the SL-PLUS™ MIA Ti/HA femoral hip stem
* is at least 21 years of age at the time of surgery
* is skeletally mature in the PI's judgment
* has consented to participate in the study by signing the EC approved ICF

Exclusion Criteria:

Patient:

* requires the use of a ceramic-on-ceramic bearing
* has infections, acute or chronic, local or systemic
* has severe muscle, nerve or vascular diseases that endanger the respective limb
* has lack of bone substance or defective bone quality that jeopardizes the stable seating of the prosthesis
* has any concomitant disease that may jeopardize implant function
* has a known allergy to study device or one or more of its components
* requires a revision surgery and has extensive bone defects
* has diagnosis of an immunosuppressive disorder
* is pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this multicenter clinical observation had at least one of the indications listed below and met all of the inclusion criteria. Patients who met any of the exclusion criteria were not eligible for this study.
  Indications:
  * Advanced hip joint wear due to degenerative, post-traumatic or rheumatoid arthritis
  * Fracture or avascular necrosis of the femoral head
  * Follow-on conditions after previous surgery such as osteosynthesis, joint reconstruction, arthrodesis, hemiarthroplasty or total hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Weymann, MD, MBA, Study Director — Smith & Nephew Orthopaedics AG
Locations (3):
- Universitätsklinik für Orthopädie, PMU Salzburg, Salzburg, Austria
- Germany (2):
  - Charité Universitätsmedizin Berlin Centrum für Muskuloskeletale Chirurgie Klinik für Orthopädie, Berlin
  - Orthopädische Chirurgie München, Munich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Unit=hips (SL-PLUS™ MIA Ti/HA stems)
Groups:
- SL-PLUS™ MIA Ti/HA: Subjects received the SL-PLUS™ MIA Ti/HA femoral hip stem and were examined using intraoperative fluoroscopic images to determine any differences between the final position of the femoral stem and the last trial rasp position. Secondarily, subjects were evaluated for leg length discrepancies preoperatively and postoperatively following insertion of the SL-PLUS™ MIA Ti/HA femoral hip stem as well as any intraoperative complications.
Period: Overall Study
Arm/Group | SL-PLUS™ MIA Ti/HA
Started | 40; 41 Unit=hips (SL-PLUS™ MIA Ti/HA stems)
Completed (There were 39 units that met the primary outcome and 41 units that met the secondary outcome.) | 38; 39 Unit=hips (SL-PLUS™ MIA Ti/HA stems)
Not Completed | 2; 2 Unit=hips (SL-PLUS™ MIA Ti/HA stems)
Not completed — Fluoroscopic images not made available | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: hips
Arm/Group | SL-PLUS™ MIA Ti/HA
Number analyzed (Participants) | 40
Number analyzed (hips) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.84 (9.393)
Sex: Female, Male [Count of Units; unit: hips]
  Female | 25
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: hips]
  Germany | 21
  Austria | 20
Operated Side [Count of Units; unit: hips]
  Left | 18
  Right | 23
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 167.68 (9.237)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 77.71 (15.837)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.47 (4.270)
Primary diagnosis for total hip arthroplasty [Count of Units; unit: hips]
  Osteoarthritis | 36
  Rheumatoid arthritis | 0
  Post-traumatic arthritis | 0
  Avascular necrosis | 2
  Dysplasia | 3
  Fracture | 0
  Other | 0
Dorr classification of femoral bone type [Count of Units; unit: hips] — Dorr Classification of femoral bone type:
  Type A: narrow canal with thick cortical walls (champagne flute canal); femoral canal width (FW)/calcar width (CW) <50%.
  Type B: moderate cortical walls; FW/CW = 50-90%.
  Type C: wide canal with thin cortical walls (stove-pipe canal); FW/CW >90%.
  The canal-to-calcar ratio is a reflection of the geometric relationship of 2 points of the proximal femoral canal. A smaller ratio represents a funnel shape and a larger ratio is a more cylindrical or stove-pipe shape.
  hips
    Type A | 3
    Type B | 32
    Type C | 6
Intraoperative used stem type [Count of Units; unit: hips]
  Standard | 34
  Lateral | 7
Intraoperative used stem size [Count of Units; unit: hips]
  Size 01 | 0
  Size 00 | 3
  Size 1 | 1
  Size 2 | 3
  Size 3 | 5
  Size 4 | 10
  Size 5 | 10
  Size 6 | 8
  Size 7 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference D Between the Position of the Last Trial Rasp and the Final Implant Position of the SL-PLUS™ MIA Ti/HA Femoral Hip Stem as Measured by an Intraoperative Fluoroscopic Measurement
Description: Difference D was measured using standardized fluoroscopic images taken during surgery. Investigators also reported any stem position corrections made as well as type of rasping instrument used.
  The difference D is given in millimeters (mm) and is defined as D = x1 - x2 with x1 being the distance between the shoulder of the trial rasp and the tip of the greater trochanter and x2 being the distance between the shoulder of the implant and the tip of the greater trochanter.
Time Frame: Intraoperative examination only
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: hips
Arm/Group | SL-PLUS™ MIA Ti/HA
Number analyzed (Participants) | 38
Number analyzed (hips) | 39
mm
  Distance X1 (trial rasp)(mm) | 7.78 [6.15 to 9.40]
  Distance X2 (stem)(mm) | 5.15 [3.52 to 6.78]
  Difference D | 2.63 [1.89 to 3.37]

2. Secondary Outcome: Number of Hips With Leg Length Discrepancy
Description: Leg length discrepancy was measured preoperatively and postoperatively shortly after insertion of the SL-PLUS™ MIA Ti/HA femoral hip stem.
Time Frame: Preoperative, directly postoperative (approximately 3 months)
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | SL-PLUS™ MIA Ti/HA
Number analyzed (Participants) | 40
Number analyzed (hips) | 41
hips
  Leg Length Discrepancy (preoperative): No Discrepancy | 24
  Leg Length Discrepancy (preoperative): Ipsilateral Longer (mm) | 1
  Leg Length Discrepancy (preoperative): Ipsilateral Shorter (mm) | 16
  Leg Length Discrepancy (postoperative): No Discrepancy | 36
  Leg Length Discrepancy (postoperative): Ipsilateral Longer (mm) | 1
  Leg Length Discrepancy (postoperative): Ipsilateral Shorter (mm) | 4

3. Secondary Outcome: Number of Hips With Intraoperative Complications
Description: Intraoperative complications were collected as a secondary outcome.
Time Frame: Intraoperative examination only
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | SL-PLUS™ MIA Ti/HA
Number analyzed (Participants) | 40
Number analyzed (hips) | 41
hips
  Adverse Events (AEs) | 0
  Serious Adverse Events (SAEs) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of preoperative examinations (Baseline) until directly postoperatively (time frame of approximately 3 months enrollment period).
Arm/Group | SL-PLUS™ MIA Ti/HA
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Basic fluoroscopic image analysis (intrinsic: resolution/technique and extrinsic: alignment/orientation to landmarks). The Guide to the Expression of Uncertainty in Measurement (GUM) was followed to estimate the combined uncertainty of the method.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator must submit results for any proposed publication to the sponsor at least 60 days before the submission. All publications will include any comments by the sponsor to modify publication for any potentially patentable item, trade secret, proprietary right, or confidential information of the sponsor. Any publication based on the results obtained from the site (or group of sites) shall not be made before the first multicenter publication.

DOCUMENTS (2):
  • Study Protocol (2015-09-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02664272/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02664272/SAP_001.pdf